CLINICAL TRIAL: NCT00756171
Title: Colesevelam Versus Placebo in Cholestatic Pruritus. A Double-blind, Placebo-controlled Study
Brief Title: Colesevelam Versus Placebo in Cholestatic Pruritus
Acronym: COPE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COPE_08
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Liver Disease
Keywords: Cholestatic; pruritus; of any cause
MeSH Terms: conditions — Pruritus | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Verum; colesevelam
  Interventions: Drug: colesevelam
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: colesevelam — 2 times 3 625 mg tablets daily, 3 weeks
  Other Names: Cholestagel
  Arms: 1
Drug: placebo — 2 times 3 625mg tablets daily
  Arms: 2

SUMMARY:
38 patients with pruritus due to chronic cholestatic liver disease will be evaluated in an investigator initiated, multicenter, double-blind, placebo-controlled, 3-week study assessing the effects of colesevelam on pruritus. Colesevelam is an oral, non-absorbable bile-acid sequestrant much more potent than cholestyramine but free of adverse effects. It is registered as a lipid lowering agent. The intensity of symptoms will be scored by means of daily Visual Analogue Scales (VAS). Fatigue, quality of life and cutaneous scratch lesions will also be evaluated using quantitative instruments.

ELIGIBILITY:
Inclusion Criteria:

* patients with pruritus as a result of a cholestatic disorder
* age above 18 years
* informed consent

Exclusion Criteria:

* use of cholestyramine
* pregnancy
* inability to understand or speak Dutch language
* malignancy/life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
40% reduction of pruritus according to visual analogue scores | 3 weeks

SECONDARY OUTCOMES:
improvement in quality of life scores | 3 weeks
Reduction in pruritus score/scratch lesions | 3 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amsterdam Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Kuiper EM, van Erpecum KJ, Beuers U, Hansen BE, Thio HB, de Man RA, Janssen HL, van Buuren HR. The potent bile acid sequestrant colesevelam is not effective in cholestatic pruritus: results of a double-blind, randomized, placebo-controlled trial. Hepatology. 2010 Oct;52(4):1334-40. doi: 10.1002/hep.23821. PMID 20683930